CLINICAL TRIAL: NCT04961424
Title: Risk Factors for Postoperative Spinal Epidural Hematoma Following Posterior Thoracic Spinal Surgery in a Single Institute
Status: Completed | Type: Observational
Sponsor: Peking University Third Hospital (Other)
Responsible Party: Principal Investigator, Li Weishi, Director of the orthopaedic department, Peking University Third Hospital
Other Study IDs: M2020006
Record Dates: First submitted 2021-06-27; First posted 2021-07-14 (Actual); Last update posted 2021-07-14 (Actual); Status verified 2021-07

CONDITIONS: Spinal Epidural Hematoma; Thoracic Surgery
Keywords: symptomatic spinal epidural hematoma; posterior thoracic surgery; local kyphosis angle; occupying ratio of cross-sectional area; cerebrospinal fluid leakage.
MeSH Terms: conditions — Hematoma, Epidural, Spinal; Cerebrospinal Fluid Leak

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Symptomatic spinal epidural hematoma Group: Patients who performed thoracic decompression surgery and developed neurological deficit after surgery due to the symptomatic spinal epidural hematoma were enrolled into case group.
- Control group: hose who did not develop the symptomatic spinal epidural hematoma, underwent the same procedures of similar complexity at the same section of thoracic spine in the same period (the same year or the following year) were randomly selected from the pool of patients.

SUMMARY:
This is a retrospective, observational single-center study. The studies is to investigate the incidence of posterior epidural spinal hematoma(PSEH) and recognize the risk factors for it in a cohort of patients undergoing posterior thoracic surgery in isolation.

DETAILED DESCRIPTION:
The study enrolled patients from January 2010 to December 2019, patients who developed PSEH after posterior thoracic surgery and underwent the hematoma evacuation. For each PSEH patients, 2 or 3 controls who did not develop the PSEH, underwent the same procedures of similar complexity at the same section of thoracic spine in the same period were collected. The preoperative and intraoperative factors, blood pressure related factors and radiographic parameters were collected to identify possible risk factors by comparing between two groups.

ELIGIBILITY:
Inclusion Criteria:

Subjects satisfying the following criteria will be considered eligible for enrollment in this study:

1. Patient is ≥ 18 years and < 80 years of age;
2. Patient who received thoracic decompression surgery via posterior approach
3. Patient who diagnosed as symptomatic spinal epidural haematoma and received revision surgery.

Exclusion Criteria:

1. Thoracic spinal stenosis caused by trauma, tumor, infectious, deformity and other disease;
2. Symptomatic spinal epidural haematoma happened at cervicothoracic and thoracolumbar junction;
3. Initial surgeries were performed at other hospital;
4. Incomplete clinical data.

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Between January 2010 and December 2019, 1612 patients were performed thoracic decompression surgery due to thoracic spinal stenosis (TSS) caused by thoracic disc herniation, ossification of posterior longitudinal ligament and ligamentum flavum with/without posterior instrumentation in our institution. The SSEH group patients were determined by symptom, MRI, intraoperative finding and underwent hematoma evacuation within one weeks of the initial surgery. For the control group, those who did not develop the SSEH, underwent the same procedures of similar complexity at the same section of thoracic spine in the same period (the same year or the following year) were randomly selected from the pool of patients.
Sampling Method: Non-Probability Sample
Enrollment: 22 (Actual)
Dates: Start 2020-02-19 (Actual); Primary Completion 2020-02-19 (Actual); Study Completion 2021-02-18 (Actual)

PRIMARY OUTCOMES:
Large local kyphosis angle | 6 months
  The local kyphosis angle was determined by the measurement of the Cobb angle. Large local kyphosis angle creates a narrow space between the paravertebral muscles and spinal cord, especially in muscles with edema after surgery. Large local kyphosis angle is considered as a risk factor for symptomatic spinal epidural hematoma
High occupying ratio of cross-sectional area | 6 months
  Severe compression on spinal epidural venous plexus lead to poor elasticity of the vessel wall and impedance of blood flow. As a result, dilatation of the spinal epidural venous plexus are more often in symptomatic spinal epidural haematoma patients, contributing to the development of haematoma. Therefore, high occupying ratio of cross-sectional area is considered as a risk factors for symptomatic spinal epidural hematoma.
Cerebrospinal fluid leakage | 6 months
  Cerebrospinal fluid leakage provides internal pressure for the dura and its own contents, and a small haematoma does not easily induce symptoms. It is the author's hypothesis that if cerebrospinal fluid leakage occurs intraoperatively, internal pressure loss, even in a small hematoma, can cause compression. Therefore, cerebrospinal fluid leakage are considered as a risk factor for symptomatic spinal epidural hematoma

CONTACTS AND LOCATIONS:
Overall Officials: Weishi Li, M.D., Principal Investigator — Peking University Third Hospital
Locations (1):
- Peking University Third hospital, Beijing, Beijing Municipality, China

IPD SHARING:
Plan to Share IPD: Yes
We will make the clinical study report available for half a year after the publication of the results of the studys
Supporting Information: CSR
Time Frame: The IPD will become available for half a year after the publication of the results of the study.
Access Criteria: The IPD is available to the readers of the journal in which our research is published. The corresponding author of the published papers will review the requests

REFERENCES:
- [Result] Leonardi MA, Zanetti M, Saupe N, Min K. Early postoperative MRI in detecting hematoma and dural compression after lumbar spinal decompression: prospective study of asymptomatic patients in comparison to patients requiring surgical revision. Eur Spine J. 2010 Dec;19(12):2216-22. doi: 10.1007/s00586-010-1483-x. Epub 2010 Jun 17. PMID 20556438
- [Result] Amiri AR, Fouyas IP, Cro S, Casey AT. Postoperative spinal epidural hematoma (SEH): incidence, risk factors, onset, and management. Spine J. 2013 Feb;13(2):134-40. doi: 10.1016/j.spinee.2012.10.028. Epub 2012 Dec 5. PMID 23218510
- [Result] Delamarter RB, Sherman J, Carr JB. Pathophysiology of spinal cord injury. Recovery after immediate and delayed decompression. J Bone Joint Surg Am. 1995 Jul;77(7):1042-9. doi: 10.2106/00004623-199507000-00010. PMID 7608226
- [Result] Yamada K, Abe Y, Satoh S, Yanagibashi Y, Hyakumachi T, Masuda T. Large Increase in Blood Pressure After Extubation and High Body Mass Index Elevate the Risk of Spinal Epidural Hematoma After Spinal Surgery. Spine (Phila Pa 1976). 2015 Jul 1;40(13):1046-52. doi: 10.1097/BRS.0000000000000876. PMID 25768686
- [Result] Fujiwara Y, Manabe H, Izumi B, Harada T, Nakanishi K, Tanaka N, Adachi N. The impact of hypertension on the occurrence of postoperative spinal epidural hematoma following single level microscopic posterior lumbar decompression surgery in a single institute. Eur Spine J. 2017 Oct;26(10):2606-2615. doi: 10.1007/s00586-017-5165-9. Epub 2017 Jun 9. PMID 28597302
- [Result] Kao FC, Tsai TT, Chen LH, Lai PL, Fu TS, Niu CC, Ho NY, Chen WJ, Chang CJ. Symptomatic epidural hematoma after lumbar decompression surgery. Eur Spine J. 2015 Feb;24(2):348-57. doi: 10.1007/s00586-014-3297-8. Epub 2014 Apr 24. PMID 24760464
- [Result] Fujita N, Michikawa T, Yagi M, Suzuki S, Tsuji O, Nagoshi N, Okada E, Tsuji T, Nakamura M, Matsumoto M, Watanabe K. Impact of lumbar hypolordosis on the incidence of symptomatic postoperative spinal epidural hematoma after decompression surgery for lumbar spinal canal stenosis. Eur Spine J. 2019 Jan;28(1):87-93. doi: 10.1007/s00586-018-5782-y. Epub 2018 Oct 9. PMID 30302540
- [Result] Knusel K, Du JY, Ren B, Kim CY, Ahn UM, Ahn NU. Symptomatic Epidural Hematoma after Elective Posterior Lumbar Decompression: Incidence, Timing, Risk Factors, and Associated Complications. HSS J. 2020 Dec;16(Suppl 2):230-237. doi: 10.1007/s11420-019-09690-2. Epub 2019 Jul 1. PMID 33380952
- [Result] Hohenberger C, Zeman F, Hohne J, Ullrich OW, Brawanski A, Schebesch KM. Symptomatic Postoperative Spinal Epidural Hematoma after Spinal Decompression Surgery: Prevalence, Risk Factors, and Functional Outcome. J Neurol Surg A Cent Eur Neurosurg. 2020 Jul;81(4):290-296. doi: 10.1055/s-0039-1697024. Epub 2020 Jan 14. PMID 31935784
- [Result] Mueller K, Altshuler M, Voyadzis JM, Sandhu FA. The incidence of symptomatic postoperative epidural hematoma after minimally invasive lumbar decompression: A single institution retrospective review. Clin Neurol Neurosurg. 2020 Aug;195:105868. doi: 10.1016/j.clineuro.2020.105868. Epub 2020 Apr 22. PMID 32361024